CLINICAL TRIAL: NCT02059239
Title: A Pilot Study of a Sequential Regimen of Intensive Chemotherapy Followed by Autologous or Allogeneic Transplantation for Refractory Lymphoma (Non-Hodgkin's and Hodgkin's) and Phase 2 Expansion Cohort
Brief Title: Bendamustine Bridge to Autologous or Allogeneic Transplant for Relapsed/Refractory Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1208012875
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Lymphoma; Transplant
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma | interventions — Bendamustine Hydrochloride; Carmustine; Etoposide; etoposide phosphate; Melphalan; Cytarabine; Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemo plus Autologous Transplantation (Experimental): Bendamustine 200 mg/ m2/ day on Days - 24 and Day - 23 followed by a short break of 10 - 14 days, followed by Melphalan, Carmustine, Etoposide, Cytarabine (BEAM) and alemtuzumab, plus rituximab for all b-cell malignancies, followed by autologous transplant
  Interventions: Drug: Bendamustine; Drug: Carmustine; Drug: Etoposide; Drug: Melphalan; Drug: Cytarabine; Drug: Alemtuzumab; Biological: Autologous Stem Cell Transplantation; Drug: Rituximab
- Chemo plus Allogeneic Transplantation (Experimental): Bendamustine 200 mg/ m2/ day on Days - 24 and Day - 23 followed by a short break of 10 - 14 days, followed by Melphalan, Carmustine, Etoposide, Cytarabine (BEAM) and alemtuzumab, plus rituximab for all b-cell malignancies, followed by allogeneic transplant
  Interventions: Drug: Bendamustine; Drug: Carmustine; Drug: Etoposide; Drug: Melphalan; Drug: Cytarabine; Drug: Alemtuzumab; Biological: Allogeneic Stem Cell Transplantation; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Days - 24 and Day - 23 followed by a short break of 10 - 14 days.
  Other Names: Treanda
Drug: Carmustine — 300 mg/m2 on Day -6
  Other Names: Bicnu
Drug: Etoposide — 100 mg/m2 on days -5 to -2
  Other Names: Etopophos; Toposar
Drug: Melphalan — 140mg/m2 on Day -1
  Other Names: Alkeran
Drug: Cytarabine — 200 mg/m2 on days -5 to -2
  Other Names: Ara-C
Drug: Alemtuzumab — 20 mg/m2 days -6 to -2 for UNRELATED donors, and 20 mg/m2 days -4 to -2 for RELATED donors
  Other Names: Campath
Biological: Autologous Stem Cell Transplantation
  Arms: Chemo plus Autologous Transplantation
Biological: Allogeneic Stem Cell Transplantation
  Arms: Chemo plus Allogeneic Transplantation
Drug: Rituximab — Only to be administered in subjects with B-cell malignancies. Dose is 375 mg/m2 on Days 1 and 8 post-transplant
  Other Names: Rituxan

SUMMARY:
This clinical trial is for men and women with whose lymphoma (non-Hodgkin or Hodgkin) did not respond to treatment or has returned after responding to previous therapy, and who are in need of a stem cell transplant.

The purpose of this study is to test the safety and effectiveness of giving the drug Bendamustine, followed by high dose chemotherapy, within two weeks prior to a stem cell transplant for lymphoma that has not achieved a complete response to salvage (treatment used for relapsed disease) chemotherapy.

DETAILED DESCRIPTION:
Subjects with Hodgkin's or Non-Hodgkin's lymphoma that did not respond to treatment or have disease that has returned after responding to previous treatment, and are in need of a stem cell transplant will be eligible for this pilot study. Thirty subjects will be enrolled, with 15 subjects assigned to the autologous transplant cohort (according to disease status and eligibility) and 15 subjects to the allogeneic transplant cohort (according to diseases status and eligibility).

Subjects will undergo the following a number of screening procedures to determine eligibility. All eligible subjects will receive bendamustine at a dose of 200 mg/ m2/ day for two days on Days - 24 and Day - 23 followed by a short break of 10 - 14 days. Subjects will then receive the conditioning regimen, BEAM (carmustine, etoposide, cytarabine arabinoside, and Melphalan) and alemtuzumab for 6 days (Day -6 to Day -1) followed by an autologous or allogeneic transplant.

Subjects with pathological confirmed B-cell malignancies will also receive rituximab 375 mg/m2 on Days + 1 and +8 post-transplant. Subjects with T-cell lymphoma will be enrolled in the study but will not receive rituximab.

After the transplantation all subjects will receive medication to prevent graft vs host disease and supportive care to prevent infections. To speed up the recovery of stem cells, subjects will receive post-transplant filgrastim (G-CSF).

After discharge from the hospital, subjects will be seen regularly in the clinic for an exam and assessments. All these tests are considered standard of care.

ELIGIBILITY:
Inclusion Criteria:

* must have histologically or cytologically confirmed relapsed or primary refractory lymphoma (including Hodgkin's Lymphoma) staged with Positron Emission Tomography (PET) scan to have

  * Allogeneic arm:

    * Progressive disease or
    * No response to salvage therapy or
    * Partial response to salvage therapy defined as > 50% reduction in bidirectional area of masses but standardized uptake value (SUV) remains ≥8 in at least some PET avid areas
    * Prior autologous transplant
  * Autologous arm:

    * Partial response of >50% reduction in bidirectional area of masses and SUV reduction to <8 in PET avid areas Subjects must have evaluable disease.
* Subjects must have received at least one induction therapy and one line of salvage therapy that each incorporate at least two drugs that are standard of care for lymphoma
* Age >18 years.
* Karnofsky Performance Score (KPS) ≥ 50%
* For autologous transplants: Subjects must have an adequate number of CD34+ stem cells collected to allow for transplantation. This number is defined as ≥ 2x106 CD34+ cells / kg body weight. If not previously collected and stored, the subject must be willing to undergo stem cell mobilization and collection as per standard practice. If sufficient cells cannot be collected, subjects will be offered the option to proceed with the allogeneic arm of the study.
* Male and female subjects must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment. Female subjects of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Known to be positive for HIV
* Subjects may not be receiving any other investigational agents (defined as non FDA-approved agents) at the time of initiating bendamustine regimen. However, the salvage therapy for lymphoma can be part of an ongoing clinical trial with an investigational agent.
* Women who are pregnant or breast feeding. Women of childbearing age must use adequate contraception and have a negative pregnancy test.
* The risks to an unborn fetus or potential risks in nursing infants are unknown.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any medications listed in the protocol.
* Subject with severely decreased Left Ventricular Ejection Fraction (LVEF) or severely impaired pulmonary function tests (PFT's)
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsiporah Shore, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Orfali N, Jhanwar Y, Koo C, Pasciolla M, Baldo M, Cuvilly E, Furman R, Gergis U, Greenberg J, Guarneri D, Hsu JM, Leonard JP, Mark T, Mayer S, Maignan K, Martin P, Opong A, Pearse R, Phillips A, Rossi A, Ruan J, Rutherford SC, Ryan J, Suhu G, Van Besien K, Shore T. Sequential intensive chemotherapy followed by autologous or allogeneic transplantation for refractory lymphoma. Leuk Lymphoma. 2021 Jul;62(7):1629-1638. doi: 10.1080/10428194.2021.1881516. Epub 2021 Feb 13. PMID 33586581

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemo Plus Autologous Transplantation: Bendamustine 200 mg/ m2/ day on Days - 24 and Day - 23 followed by a short break of 10 - 14 days, followed by Melphalan, Carmustine, Etoposide, Cytarabine (BEAM) and alemtuzumab, plus rituximab for all b-cell malignancies, followed by autologous transplant
  Bendamustine: Days - 24 and Day - 23 followed by a short break of 10 - 14 days.
  Carmustine: 300 mg/m2 on Day -6
  Etoposide: 100 mg/m2 on days -5 to -2
  Melphalan: 140mg/m2 on Day -1
  Cytarabine: 200 mg/m2 on days -5 to -2
  Alemtuzumab: 20 mg/m2 days -6 to -2 for UNRELATED donors, and 20 mg/m2 days -4 to -2 for RELATED donors
  Autologous Stem Cell Transplantation
  Rituximab: Only to be administered in subjects with B-cell malignancies. Dose is 375 mg/m2 on Days 1 and 8 post-transplant
- Chemo Plus Allogeneic Transplantation: Bendamustine 200 mg/ m2/ day on Days - 24 and Day - 23 followed by a short break of 10 - 14 days, followed by Melphalan, Carmustine, Etoposide, Cytarabine (BEAM) and alemtuzumab, plus rituximab for all b-cell malignancies, followed by allogeneic transplant
  Bendamustine: Days - 24 and Day - 23 followed by a short break of 10 - 14 days.
  Carmustine: 300 mg/m2 on Day -6
  Etoposide: 100 mg/m2 on days -5 to -2
  Melphalan: 140mg/m2 on Day -1
  Cytarabine: 200 mg/m2 on days -5 to -2
  Alemtuzumab: 20 mg/m2 days -6 to -2 for UNRELATED donors, and 20 mg/m2 days -4 to -2 for RELATED donors
  Allogeneic Stem Cell Transplantation
  Rituximab: Only to be administered in subjects with B-cell malignancies. Dose is 375 mg/m2 on Days 1 and 8 post-transplant
Period: Overall Study
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Started | 18 | 16
Completed | 16 | 13
Not Completed | 2 | 3
Not completed — Progressive Disease after Bendamustine | 1 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 12 | 9 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34
Diagnosis [Count of Participants; unit: Participants]
  Diffuse Large B-Cell Lymphoma | 6 | 1 | 7
  Follicular Lymphoma | 2 | 1 | 3
  Hodgkin's Disease | 5 | 3 | 8
  Mantle Cell Lymphoma | 2 | 1 | 3
  Transformed Diffuse Large B-Cell Lymphoma | 2 | 4 | 6
  Peripheral T-Cell Lymphoma | 0 | 2 | 2
  Other | 1 | 4 | 5
Lines of Prior Therapy [Number; unit: Lines of Therapy]
  2 Lines | 11 | 3 | 14
  3 Lines | 4 | 3 | 7
  4 Lines | 1 | 5 | 6
  5+ Lines | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Able to Proceed to Transplant
Description: Number of patients in each arm able to proceed to stem cell transplantation within 14 days of receiving bendamustine treatment
Time Frame: 14 days after bendamustine treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 18 | 16
Participants
  Proceeded to Transplant | 16 | 13
  Did Not Proceed to Transplant - Physician Decision | 1 | 0
  Did Not Proceed to Transplant - Progressive Disease | 1 | 3
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 88.9, 95% CI 2-sided [65.3 to 98.6]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 81.3, 95% CI 2-sided [54.4 to 95.9]

2. Primary Outcome: Number of Patients Achieving Neutrophil Engraftment
Description: Proportion of patients who successfully achieve neutrophil engraftment after stem cell transplant, defined as an absolute neutrophil count of 500/mm3 or for three consecutive days.
Time Frame: 35 Days Post-Transplant
Population: 5 participants (2 from chemo + autologous transplant arm, 3 from chemo + allogeneic transplant arm) were unable to be analyzed for this outcome measure as they did not complete the study and did not receive an autologous or allogeneic transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 16 | 13
Participants | 16 | 13
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 100.0, 95% CI 2-sided [79.4 to 100.0]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 100.0, 95% CI 2-sided [75.3 to 100.0]

3. Primary Outcome: Number of Patients Achieving Platelet Engraftment
Description: Proportion of patients who successfully achieve platelet engraftment after stem cell transplant, defined as a platelet count of >20k/microL for three consecutive days without transfusion support for seven consecutive days.
Time Frame: 74 Days Post-Transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 16 | 13
Participants | 16 | 12
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 100.0, 95% CI 2-sided [79.4 to 100.0]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 92.3, 95% CI 2-sided [64.0 to 99.8]

4. Secondary Outcome: Overall Survival at Day 100 Post-Transplant
Description: The time from stem cell infusion (Day 0) to death from any cause.
Time Frame: From Day 0 until time of death, assessed up to 100 days post-transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 16 | 13
Participants
  Alive | 16 | 11
  Deceased | 0 | 2
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 100.0, 95% CI 2-sided [79.4 to 100.0]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 84.6, 95% CI 2-sided [54.6 to 98.1]

5. Secondary Outcome: Overall Survival at Day 365 Post-Transplant
Description: The time from stem cell infusion (Day 0) to death from any cause.
Time Frame: From Day 0 until time of death, assessed up to 365 days post-transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 16 | 13
Participants
  Alive | 16 | 6
  Deceased | 0 | 7
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 100.0, 95% CI 2-sided [79.4 to 100.0]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 46.2, 95% CI 2-sided [19.2 to 74.9]

6. Secondary Outcome: Transplant-Related Mortality
Description: Death due to any cause other than disease progression within first 100 days post-transplant.
Time Frame: From Day 0 until time of death, up to 100 days post-transplant.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 16 | 13
Participants | 0 | 2
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 0.0, 95% CI 2-sided [0.0 to 20.6]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 15.4, 95% CI 2-sided [1.9 to 45.4]

7. Secondary Outcome: Disease Response Following Salvage Chemotherapy
Description: Proportion of patients achieving a complete remission (CR; disappearance of clinically overt disease with no FDG-avid lesions on PET scan), partial remission (PR; reduction in clinical disease buden and >50% bi-dimensional decrease in tumor size on imaging), stable disease (SD; failure to meet the criteria for CR, PR or PD with no new areas of disease involvement) or progressive disease (PD; the appearance of any new lesion >1.5cm in size or a greater than 50% increase in the diameter of a previously identified node of over 1cm in size), as per Cheson Criteria, following salvage chemotherapy with Bendamustine.
Time Frame: Within 14 days of salvage chemotherapy treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 18 | 16
Participants
  Complete Remission | 4 | 1
  Partial Remission | 8 | 6
  Stable Disease | 4 | 2
  Progressive Disease | 1 | 6
  Not Assessed | 1 | 1
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion (objective response: CR+PR) in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 66.7, 95% CI 2-sided [41.0 to 86.7]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion (objective response: CR+PR) in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 43.8, 95% CI 2-sided [19.8 to 70.1]

8. Secondary Outcome: Disease Response 30 Days Post-Transplant
Description: Proportion of patients achieving a complete remission (CR; disappearance of clinically overt disease with no FDG-avid lesions on PET scan), partial remission (PR; reduction in clinical disease buden and >50% bi-dimensional decrease in tumor size on imaging), stable disease (SD; failure to meet the criteria for CR, PR or PD with no new areas of disease involvement) or progressive disease (PD; the appearance of any new lesion >1.5cm in size or a greater than 50% increase in the diameter of a previously identified node of over 1cm in size), as per Cheson Criteria, 30 days following autologous or allogeneic stem cell transplant
Time Frame: 30 days after stem cell transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 16 | 13
Participants
  Complete Remission | 12 | 7
  Partial Remission | 2 | 3
  Stable Disease | 2 | 1
  Progressive Disease | 0 | 1
  Not Assessed | 0 | 1
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion (objective response: CR+PR) in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 87.5, 95% CI 2-sided [61.7 to 98.4]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion (objective response: CR+PR) in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 76.9, 95% CI 2-sided [46.2 to 95.0]

9. Secondary Outcome: Disease Response at 1 Year Post-Transplant
Description: Proportion of patients achieving a complete remission (CR; disappearance of clinically overt disease with no FDG-avid lesions on PET scan), partial remission (PR; reduction in clinical disease buden and >50% bi-dimensional decrease in tumor size on imaging), stable disease (SD; failure to meet the criteria for CR, PR or PD with no new areas of disease involvement) or progressive disease (PD; the appearance of any new lesion >1.5cm in size or a greater than 50% increase in the diameter of a previously identified node of over 1cm in size), as per Cheson Criteria, 1 year following autologous or allogeneic stem cell transplant
Time Frame: 1 year after stem cell transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 16 | 13
Participants
  Complete Remission | 12 | 4
  Partial Remission | 1 | 0
  Stable Disease | 0 | 0
  Progressive Disease | 3 | 2
  Not Assessed | 0 | 0
  Patient Deceased | 0 | 7
Statistical Analysis 1: Comparison: Chemo Plus Autologous Transplantation; Test type: Other — Simple proportion (objective response: CR+PR) in autologous group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 81.3, 95% CI 2-sided [54.4 to 96.0]
Statistical Analysis 2: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Simple proportion (objective response: CR+PR) in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Proportion (percent) = 30.8, 95% CI 2-sided [9.1 to 61.4]

10. Secondary Outcome: Progression-Free Survival After Stem Cell Transplant
Description: Time elapsed between stem cell transplant (Day 0) and disease progression, as defined by the Cheson Criteria (the appearance of any new lesion >1.5cm in size or a greater than 50% increase in the diameter of a previously identified node of over 1cm in size)
Time Frame: Stem cell transplant (Day 0) up to 2 years post-transplant
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemo Plus Autologous Transplantation | Chemo Plus Allogeneic Transplantation
Number analyzed (Participants) | 16 | 13
Months | NA [NA to NA] — Median progression-free survival was not reached in the chemo plus autologous transplantation group. An insufficient number of patients experienced progression/death within the follow-up interval to enable calculation of the median and both the upper and lower limits of the 95% confidence interval. | 8 [5 to 25]
Statistical Analysis 1: Comparison: Chemo Plus Allogeneic Transplantation; Test type: Other — Median PFS in allogeneic group with exact (Clopper-Pearson) 95% confidence interval; Median (95% CI) = 8, 95% CI 2-sided [5 to 25]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed Day -24 (start of Bendamustine treatment) through 1 year post-transplant.
Description: All adverse events were first documented by the study transplant physicians and thereafter collated and graded by two independent reviewed according to CTCAE version 4.0. 5 participants (2 autologous, 3 allogeneic) did not proceed to transplant and were not evaluable for adverse events on the Chemo Plus Autologous Transplant or Chemo Plus Allogeneic Transplant arms.
Groups:
- Bendamustine: Bendamustine 200 mg/ m2/ day on Days - 24 and Day - 23 followed by a short break of 10 - 14 days
- Bendamustine Plus Autologous Transplantation: Bendamustine 200 mg/ m2/ day on Days - 24 and Day - 23 followed by a short break of 10 - 14 days, followed by Melphalan, Carmustine, Etoposide, Cytarabine (BEAM) and alemtuzumab, plus rituximab for all b-cell malignancies, followed by autologous transplant
  Bendamustine: Days - 24 and Day - 23 followed by a short break of 10 - 14 days.
  Carmustine: 300 mg/m2 on Day -6
  Etoposide: 100 mg/m2 on days -5 to -2
  Melphalan: 140mg/m2 on Day -1
  Cytarabine: 200 mg/m2 on days -5 to -2
  Alemtuzumab: 20 mg/m2 days -6 to -2 for UNRELATED donors, and 20 mg/m2 days -4 to -2 for RELATED donors
  Autologous Stem Cell Transplantation
  Rituximab: Only to be administered in subjects with B-cell malignancies. Dose is 375 mg/m2 on Days 1 and 8 post-transplant
- Bendamustine Plus Allogeneic Transplantation: Bendamustine 200 mg/ m2/ day on Days - 24 and Day - 23 followed by a short break of 10 - 14 days, followed by Melphalan, Carmustine, Etoposide, Cytarabine (BEAM) and alemtuzumab, plus rituximab for all b-cell malignancies, followed by allogeneic transplant
  Bendamustine: Days - 24 and Day - 23 followed by a short break of 10 - 14 days.
  Carmustine: 300 mg/m2 on Day -6
  Etoposide: 100 mg/m2 on days -5 to -2
  Melphalan: 140mg/m2 on Day -1
  Cytarabine: 200 mg/m2 on days -5 to -2
  Alemtuzumab: 20 mg/m2 days -6 to -2 for UNRELATED donors, and 20 mg/m2 days -4 to -2 for RELATED donors
  Allogeneic Stem Cell Transplantation
  Rituximab: Only to be administered in subjects with B-cell malignancies. Dose is 375 mg/m2 on Days 1 and 8 post-transplant
Arm/Group | Bendamustine | Bendamustine Plus Autologous Transplantation | Bendamustine Plus Allogeneic Transplantation
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/16 | 7/13
Serious Adverse Events (participants affected / at risk) | 2/34 | 4/16 | 10/13
Other Adverse Events (participants affected / at risk) | 9/34 | 16/16 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=34) | Bendamustine Plus Autologous Transplantation (N=16) | Bendamustine Plus Allogeneic Transplantation (N=13)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Intestinal Necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Disseminated Adenovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post-Transplant Lymphoproliferative Disorder (Investigations) | 0 (0) | 0 (0) | 2 (2)
Chronic Graft versus Host Disease (Investigations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Acute Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
Myelodysplastic Syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Myeloid Leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=34) | Bendamustine Plus Autologous Transplantation (N=16) | Bendamustine Plus Allogeneic Transplantation (N=13)
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 11 (11) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Oral Mucositis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Cytomegalovirus Viremia (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Epstein-Barr Virus Viremia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Lung Infection - Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Lung Infection - Viral Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung Infection - Fungal Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 13 (14)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Norovirus Enterocolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection - Influenza A (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection - Rhinovirus (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper Respiratory Infection - Respiratory Syncytial Virus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT02059239/Prot_SAP_000.pdf